CLINICAL TRIAL: NCT03101150
Title: Effect of Antenatal Vitamin D3 Supplementation on Risk of Pre-eclampsia
Brief Title: Effect of Vitamin D3 Supplementation in Pregnancy on Risk of Pre-eclampsia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Aisha Mansoor Ali, Assistant Consultant Obstetric and Gynecology, King Fahad Medical City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00008644
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-02

CONDITIONS: Vitamin D Deficiency; Pre-Eclampsia
Keywords: Maternal vitamin D; Deficiency; Insufficiency; Pregnancy; Pre-eclampsia; IUGR
MeSH Terms: conditions — Vitamin D Deficiency; Pre-Eclampsia | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 400 IU Vitamin D3 (Active Comparator): 400IU vitamin D3 contained in antenatal multivitamin once daily by mouth starting from 14 weeks of pregnancy till delivery.
  Interventions: Drug: 400 IU Vitamin D3
- 4000 IU Vitamin D3 (Experimental): 4000 IU Vitamin D3 drops once daily by mouth starting from 14 weeks of pregnancy till delivery.
  Interventions: Drug: 4000 IU Vitamin D3

INTERVENTIONS:
Drug: 400 IU Vitamin D3 — Antenatal multivitamin
  Other Names: Materna
  Arms: 400 IU Vitamin D3
Drug: 4000 IU Vitamin D3 — 4000 IU Vitamin D3 (cholecalciferol) daily = 40 drops daily
  Other Names: Vidrop
  Arms: 4000 IU Vitamin D3

SUMMARY:
Vitamin D deficient pregnant ladies were selected and randomized into 2 groups for routine daily dose of multivitamin (400IU vitamin D3) versus maximum safest treatment daily dose (4000IU vitamin D3). Participants were assessed and compared for number of pre-eclampsia cases.

DETAILED DESCRIPTION:
Vitamin D3 has key role in decidualization and implantation of placenta.Vitamin D deficiency is thought to have positive association with pre-eclampsia.Vitamin D deficiency is highly prevalent in some parts of the world and it is not universally screened antenatally. Pre-eclampsia is a known multifactorial pregnancy disorder with significant maternal and perinatal morbidity and mortality. Vitamin D3 has a down-regulating effect on inflammatory pathways and reducing endothelial cell damage.

Investigators want to assess in vitamin D deficient group whether treatment reduces the risk of pre-eclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed singleton pregnancy of less than 13 completed weeks of gestation at the time of consent.
* Planned to receive antenatal care in King Fahad Medical City antenatal clinic.
* The ability to provide written informed consent at the first visit.
* Low risk pregnancy; and Serum vitamin D3 levels less than < 25nmol/L.

Exclusion Criteria:

* Mothers with pregnancy with abnormal foetus.
* Previous history of hypertension, pre-eclampsia, recurrent miscarriages.
* Chronic kidney disease, chronic liver disease, and malignancy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant population
Enrollment: 179 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2015-12-31 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 416 participants were screened. 192 did not meet eligibility criteria. 38 refused to participate and 7 turned out to be ectopic pregnancy.
Groups:
- 400 IU: Materna tablet once daily orally from 14 weeks of pregnancy til delivery.
- 4000 IU: Vidrop vitamin D 40 drops daily orally from 14 weeks of pregnancy till delivery.
Period: Overall Study
Arm/Group | 400 IU | 4000 IU
Started | 86 | 93
Completed | 81 | 83
Not Completed | 5 | 10
Not completed — Lost to Follow-up | 2 | 4
Not completed — Miscarriage | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 IU Vitamin D3 | 4000 IU Vitamin D3 | Total
Number analyzed (Participants) | 86 | 93 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (5.3) | 29.4 (4.8) | 29.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 93 | 179
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Saudi Arabia | 80 | 80 | 160
  India | 3 | 5 | 8
  Philippines | 3 | 7 | 10
  Africa | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 28.8 (7.3) | 28.1 (7.2) | 28.4 (7.2)
Primiparity [Count of Participants; unit: Participants] | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pre-eclampsia in Both Arms
Description: Occurrence of pre-eclampsia or not in all patients irrespective of Vitamin D dose.
Time Frame: From 20 weeks of pregnancy till event of pre-eclampsia seen, whichever came first, assessed up to 32 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | 400 IU | 4000 IU
Number analyzed (Participants) | 81 | 83
Participants | 6 | 1
Statistical Analysis 1: Comparison: 400 IU vs 4000 IU; Eligible and consented study subjects were randomized according to permuted block design scheme to be allocated in 400 IU arm and 4000 IU arm; Test type: Other — A sample size of minimum 152 was calculated to be able to determine incidence of preeclampsia that is in the range of 8-17% with 80% power assuming an alpha of 5%; p < 0.05, Chi-squared; Risk Ratio (RR) = 0.163, 95% CI 2-sided [0.02 to 1.32]

2. Secondary Outcome: Change in Vitamin D Level
Description: Level of Improvement in Vitamin D status in both arms
Time Frame: At 36th week of pregnancy
Population: Out of 86 participants randomized for the arm of 400 IU, 3 had miscarriage and 2 lost to follow. So 81 participants were analyzed.
  Out of 93 participants randomized for the arm of 4000 IU, 6 had miscarriage and 4 lost to follow. So 83 were analyzed in that arm.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | 400 IU | 4000 IU
Number analyzed (Participants) | 81 | 83
nmol/L | 35.3 (20.7) | 72.3 (30.9)
Statistical Analysis 1: Comparison: 400 IU vs 4000 IU; Test type: Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Number of Patients With Intrauterine Growth Retardation
Description: Patients having fetus with retardation of growth in both arms.
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 400 IU | 4000 IU
Number analyzed (Participants) | 81 | 83
Participants | 18 | 8
Statistical Analysis 1: Comparison: 400 IU vs 4000 IU; Test type: Other; p < 0.02, Chi-squared; Risk Ratio (RR) = 0.43, 95% CI 2-sided [0.19 to 0.94]

ADVERSE EVENTS:
Arm/Group | 400 IU | 4000 IU
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/93
Other Adverse Events (participants affected / at risk) | 0/86 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes